CLINICAL TRIAL: NCT01088438
Title: Measuring Quality of Medical Student Performance at Contextualizing Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: The National Board of Medical Examiners (Other)
Responsible Party: Alan Schwartz, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: NBME0708-12
Record Dates: First submitted 2010-03-12; First posted 2010-03-17 (Estimated); Results first posted 2011-05-06 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2011-03

CONDITIONS: Education, Medical, Undergraduate; Medical History Taking; Diagnosis
Keywords: medical education; decision making; diagnostic error; contextualization
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contextualization workshop (Experimental): A four-hour course on contextualization.
  Interventions: Behavioral: Contextualization workshop
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Contextualization workshop — A four-hour course on contextualization.
  Arms: Contextualization workshop

SUMMARY:
During the project, fourth-year medical students participating in a Medicine sub-internship will be randomized to an intervention group or a control group; the intervention group will receive additional training in the application of qualitative methodology to elicit and incorporate contextual factors in the clinical encounter. All students will participate in an SP assessment consisting of four standardized patients (SPs), blinded to trial arm, presenting cases with and without important biomedical and contextual factors in a counterbalanced factorial design. Performance will be compared between trial arms; the investigators hypothesize better performance in the intervention arm. In addition, performance will be compared with United States Medical Licensing Exam (USMLE) Step 2 clinical knowledge scores to determine whether contextualizing ability is independent of clinical knowledge, and consistency of performance across individual SP cases will be studied to determine the number of cases necessary to achieve sufficient reliability for the assessment to be used.

DETAILED DESCRIPTION:
Clinical decision making requires two distinct skills: the ability to classify patients' conditions into diagnostic and management categories that permit the application of "best evidence" guidelines, and the ability to individualize or - more precisely - to contextualize care for patients whose circumstances and needs require variation from the standard approach to care. Most assessment in medical education places heavy emphasis on biomedical decision-making with little emphasis on how to incorporate contextual factors that may be essential to planning patients' care.

The goal of this project is to demonstrate and provide validity evidence for an innovative standardized patient (SP) method of assessing medical students in the clinical years on their ability to detect and respond to individual contextual factors in a patient encounter that overcomes the aforementioned challenges.

During the project, fourth-year medical students participating in a Medicine sub-internship will be randomized to an intervention group or a control group; the intervention group will receive additional training in the application of qualitative methodology to elicit and incorporate contextual factors in the clinical encounter. All students will participate in an SP assessment consisting of four SPs, blinded to trial arm, presenting cases with and without important biomedical and contextual factors in a counterbalanced factorial design. Performance will be compared between trial arms. In addition, performance will be compared with United States Medical Licensing Exam (USMLE) Step 2 clinical knowledge scores to determine whether contextualizing ability is independent of clinical knowledge, and consistency of performance across individual SP cases will be studied to determine the number of cases necessary to achieve sufficient reliability for the assessment to be used.

ELIGIBILITY:
Inclusion Criteria:

* Fourth-year medical students at University of Illinois at Chicago

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2008-07; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Schwartz, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Result] Schwartz A, Weiner SJ, Harris IB, Binns-Calvey A. An educational intervention for contextualizing patient care and medical students' abilities to probe for contextual issues in simulated patients. JAMA. 2010 Sep 15;304(11):1191-7. doi: 10.1001/jama.2010.1297. PMID 20841532

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All fourth-year medical students at the University of Illinois at Chicago (UIC) College of Medicine who were enrolled in internal medicine subinternships at one of 2 sites (UIC or Jesse Brown Veterans Administration Medical Center) July 2008 - April 2009 or August 2009 - April 2010 were eligible.
Period: Overall Study
Arm/Group | Contextualization Workshop | Control
Started | 94 | 95
Completed | 65 | 59
Not Completed | 29 | 36
Not completed — Withdrawal by Subject | 11 | 6
Not completed — Lost to Follow-up | 18 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Contextualization Workshop | Control | Total
Number analyzed (Participants) | 94 | 95 | 189
Age Continuous [Mean (Standard Deviation); unit: years] | 28.8 (3.6) | 28.8 (3.6) | 28.8 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 41 | 90
  Male | 45 | 54 | 99
Race/Ethnicity, Customized [Number; unit: participants] — Number of participants identifying as "White" race.
  participants
    White | 30 | 34 | 64
    Non-White | 64 | 61 | 125

OUTCOME MEASURES:

1. Primary Outcome: Developing an Appropriate Treatment Plan (for Contextual Variant of Encounters)
Description: Probability that the learner writes a correct treatment plan for the standardized patient encounters undertaken at assessment at end of subinternship that include contextual red flags. All learners are scheduled to see 4 encounters, based on combinations of four cases and four potential variants (baseline, biomedical, contextual, biocontextual) with counterbalancing by study month; each has a single contextual variant encounter. Treatment plans are assessed by an investigator blinded to the learner's assignment to intervention or control group.
Time Frame: 1 month
Population: ITT. In one case, a participant did not receive a contextual variant encounter because the standardized patient was ill, and this encounter is excluded.
Measure: Number (95% Confidence Interval); unit: proportion of contextual encounters
Units Other Than Participants: encounters (contextual variant)
Arm/Group | Contextualization Workshop | Control
Number analyzed (Participants) | 65 | 59
Number analyzed (encounters (contextual variant)) | 64 | 59
proportion of contextual encounters | 0.67 [0.55 to 0.79] | 0.24 [0.13 to 0.35]
Statistical Analysis 1: Comparison: Contextualization Workshop vs Control; Null hypothesis: proportion of encounters with contextual red flag in which appropriate treatment is planned is the same in the two groups; Test type: Superiority or Other; p < 0.001, Chi-squared; 1 degree of freedom

2. Primary Outcome: Probing for Contextual Issues
Description: Probability that the learner probes contextual red flags raised in standardized patient encounters undertaken at assessment at end of subinternship. Each learner undertakes four encounters, each of which presents a contextual red flag that may or may not be probed; in a small number of cases, the standardized patient was ill and the learner undertook fewer than four encounters as a result. Assessment of probing is made by an investigator blinded to learner's assignment to group.
Time Frame: 1 month
Population: ITT
Measure: Number (95% Confidence Interval); unit: proportion of encounters
Units Other Than Participants: encounters
Arm/Group | Contextualization Workshop | Control
Number analyzed (Participants) | 65 | 59
Number analyzed (encounters) | 258 | 236
proportion of encounters | 0.86 [0.82 to 0.90] | 0.61 [0.55 to 0.67]
Statistical Analysis 1: Comparison: Contextualization Workshop vs Control; Null hypothesis is equal proportion of contextual red flags probed in control and intervention groups; Test type: Superiority or Other; p < .001, Chi-squared; 1 degree of freedom

3. Primary Outcome: Probing for Biomedical Issues
Description: Probability that the learner probes biomedical red flags raised in standardized patient encounters undertaken at assessment at end of subinternship. Each learner undertakes four encounters, each of which presents a biomedical red flag that may or may not be probed; in a small number of cases, the standardized patient was ill and the learner undertook fewer than four encounters as a result. Assessment of probing is made by an investigator blinded to learner's assignment to group.
Time Frame: 1 month
Population: ITT
Measure: Number (95% Confidence Interval); unit: proportion of encounters
Units Other Than Participants: encounters
Arm/Group | Contextualization Workshop | Control
Number analyzed (Participants) | 65 | 59
Number analyzed (encounters) | 258 | 236
proportion of encounters | 0.77 [0.72 to 0.82] | 0.77 [0.72 to 0.82]
Statistical Analysis 1: Comparison: Contextualization Workshop vs Control; Null hypothesis is equal proportion of encounters probed in control and intervention groups; Test type: Superiority or Other; p = 0.85, Chi-squared; 1 df

ADVERSE EVENTS:
Arm/Group | Contextualization Workshop | Control
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/95
Other Adverse Events (participants affected / at risk) | 0/94 | 0/95

LIMITATIONS AND CAVEATS:
Small number of cases and variants. Alternating assignment of site to intervention/control. Substantial drop-out (sensitivity analysis finds results robust to conservative imputation for drop-outs).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No